CLINICAL TRIAL: NCT03959436
Title: Prospective Observational Database Evaluating Outcomes of Using Carbetocin (Duratocin®) as the Primary Uterotonic Following Cesarean Delivery at Maisonneuve-Rosemont Hospital
Brief Title: Database Evaluating Outcomes of Using Carbetocin as the Primary Uterotonic Following Cesarean Delivery
Status: Completed | Type: Observational
Sponsor: Maisonneuve-Rosemont Hospital (Other)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, Valerie Zaphiratos, Unit Chief of Obstetric Anesthesia, Maisonneuve-Rosemont Hospital
Other Study IDs: 2017-836
Record Dates: First submitted 2019-05-20; First posted 2019-05-22 (Actual); Last update posted 2019-05-29 (Actual); Status verified 2019-05

CONDITIONS: Carbetocin; Cesarean Section Complications; Uterotonics; Uterine Atony With Hemorrhage
MeSH Terms: interventions — carbetocin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Carbetocin — Carbetocin as the primary uterotonic for all cesarean sections
  Other Names: Duratocin

SUMMARY:
Carbetocin (Duratocin®) is a long-acting form of oxytocin, with a half-life almost 10 times longer. Studies have demonstrated that carbetocin diminishes the need for secondary uterotonic agents compared to oxytocin for cesarean delivery (CD). Despite certain Canadian guidelines recommending its use for elective CD, several Canadian centers and other countries have not adopted carbetocin. The purpose of this study is to prospectively gather electronic data on all CDs over a one year period, elective and emergent, in a single institution, and to evaluate the efficacy and other clinical outcomes when carbetocin is used as a first line uterotonic for all CDs. A database using Microsoft Dynamics CRM is available on smart phones and tablets. Data regarding additional uterotonic use and impact of carbetocin use during CD on intra and postoperative outcomes are gathered and analyzed. The primary outcome is the use of additional uterotonics in this population compared to that described in the literature for oxytocin as the primary uterotonic.

ELIGIBILITY:
Inclusion Criteria:

* All Cesarean deliveries in the operating room.

Exclusion Criteria:

* Vaginal deliveries and double set-up vaginal deliveries conducted in the operating room.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Pregnant patients requiring cesarean section.
Sampling Method: Probability Sample
Enrollment: 612 (Actual)
Dates: Start 2017-03-29 (Actual); Primary Completion 2018-03-16 (Actual); Study Completion 2018-03-16 (Actual)

PRIMARY OUTCOMES:
Use of additional uterotonics | 24 hours
  The number of participants requiring additional uterotonics after using carbetocin as the initial uterotonic

CONTACTS AND LOCATIONS:
Overall Officials: Valerie Zaphiratos, MSc, MD, Principal Investigator — Maisonneuve-Rosemont Hospital; Philippe Richebé, MD, PhD, Principal Investigator — Maisonneuve-Rosemont Hospital
Locations (1):
- Maisonneuve-Rosemont hospital, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: Yes
To publish this data in a journal. Data includes primary outcomes and secondary outcomes related to uterotonic use and uterine atony and hemorrhage.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Our plan is to publish in the coming year.

REFERENCES:
- [Background] Boucher M, Horbay GL, Griffin P, Deschamps Y, Desjardins C, Schulz M, Wassenaar W. Double-blind, randomized comparison of the effect of carbetocin and oxytocin on intraoperative blood loss and uterine tone of patients undergoing cesarean section. J Perinatol. 1998 May-Jun;18(3):202-7. PMID 9659650
- [Background] Dansereau J, Joshi AK, Helewa ME, Doran TA, Lange IR, Luther ER, Farine D, Schulz ML, Horbay GL, Griffin P, Wassenaar W. Double-blind comparison of carbetocin versus oxytocin in prevention of uterine atony after cesarean section. Am J Obstet Gynecol. 1999 Mar;180(3 Pt 1):670-6. doi: 10.1016/s0002-9378(99)70271-1. PMID 10076146
- [Background] Borruto F, Treisser A, Comparetto C. Utilization of carbetocin for prevention of postpartum hemorrhage after cesarean section: a randomized clinical trial. Arch Gynecol Obstet. 2009 Nov;280(5):707-12. doi: 10.1007/s00404-009-0973-8. Epub 2009 Feb 20. PMID 19229549
- [Background] Attilakos G, Psaroudakis D, Ash J, Buchanan R, Winter C, Donald F, Hunt LP, Draycott T. Carbetocin versus oxytocin for the prevention of postpartum haemorrhage following caesarean section: the results of a double-blind randomised trial. BJOG. 2010 Jul;117(8):929-36. doi: 10.1111/j.1471-0528.2010.02585.x. Epub 2010 May 19. PMID 20482535
- [Background] Leduc D, Senikas V, Lalonde AB; CLINICAL PRACTICE OBSTETRICS COMMITTEE. Active management of the third stage of labour: prevention and treatment of postpartum hemorrhage. J Obstet Gynaecol Can. 2009 Oct;31(10):980-993. doi: 10.1016/S1701-2163(16)34329-8. PMID 19941729
- [Background] Su LL, Chong YS, Samuel M. Carbetocin for preventing postpartum haemorrhage. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD005457. doi: 10.1002/14651858.CD005457.pub4. PMID 22513931